CLINICAL TRIAL: NCT04957368
Title: Sustained Mood Improvement With Laughing Gas Exposure: A Randomized Controlled Pilot Trial
Acronym: SMILE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 21-096
Record Dates: First submitted 2021-04-26; First posted 2021-07-12 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder
Keywords: Feasibility trial; Nitrous Oxide
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Oxygen; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrous Oxide + saline solution (Experimental)
  Interventions: Drug: Nitrous Oxide 99 %
- Oxygen + Midazolam (Active Comparator)
  Interventions: Drug: Oxygen + Midazolam

INTERVENTIONS:
Drug: Nitrous Oxide 99 % — Nitrous oxide will be administered at an inspiratory concentration of 50% with concurrent intravenous saline (100ml) for one hour.
  Arms: Nitrous Oxide + saline solution
Drug: Oxygen + Midazolam — Oxygen will be administered at 50% with intravenous midazolam (0.02mg/kg in 100ml) for one hour
  Arms: Oxygen + Midazolam

SUMMARY:
The purpose of the study is to investigate a short-term treatment option for major depressive disorders by administering nitrous oxide gas. At this time, the main purpose is to complete a feasibility study with 40 participants suffering from treatment-resistant depression. Participants will be randomized to (1) Study group: Nitrous oxide (inhaled) + solution of saline (injected) and the (2) Control group: Oxygen (inhaled) + Midazolam (injected) as an Active Placebo.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years of age
2. Meeting Diagnostic and Statistical Manual for Mental Disorders (DSM-5) criteria for Major Depressive Disorder (MDD)
3. Current major depressive episode as confirmed by the Mini International Neuropsychiatric Interview (MINI) for DSM-5
4. Experiencing moderate to severe depressive episode, as defined by the Hamilton Depression Rating Scale (HAMD)>17
5. Failure of two trials of antidepressant therapy of adequate dose and duration, during the current depressive episode
6. For women of childbearing potential, use of highly effective or double-barrier methods of contraception. Abstinence is acceptable if it is the preferred and usual lifestyle of the female participant
7. Capacity to provide informed consent.

Exclusion criteria

1. Acute suicidality defined as score ≥3 on HAMD item 3
2. Major Depressive Episode in people with Bipolar Disorder
3. Current substance abuse or dependence and/or history of alcohol abuse or dependence within the past year
4. Dementia
5. Current or lifetime history of schizophrenia or schizoaffective disorder
6. Current history of dissociative disorders
7. Known history of hypersensitivity or allergy to Nitrous Oxide, Midazolam or any ingredients in the study formulations
8. Contraindication to receiving nitrous oxide
9. Chronic cobalamin or folate deficiency
10. Contraindication to receiving the placebo midazolam
11. Use of centrally acting medicinal products, such as opioid agonists, morphine derivatives, benzodiazepines and/or other central nervous system depressants such as barbiturates and alcohol
12. Pregnancy or breastfeeding in female participants
13. Electroconvulsive therapy within the current depressive episode
14. Receiving ketamine treatment within the current depressive episode
15. Unwilling to maintain current antidepressant regimen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 2 Years
  Recruitment rate
Withdrawal rate | 2 Years
Adherence rate | 2 Years
  Feasibility
Frequency of adverse events | 2 Years
  Safety and tolerability

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRAS) Score 0-60 (Higher scores represent higher depression). Measure changes in symptoms of depression | 6 weeks
  Frequencies on numbers of 1.- Remissions (defined as MADRS score < 10), 2.- Responses (defined as ≥ 50% reduction in MADRS score from baseline) 3.- No Responses
Toronto Side Effects Scale (TSES) - 32 items (each item has a score 1-25; higher score means higher intensity). Measure adverse side effects from antidepressant treatment | 6 weeks
  Frequencies of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No individual participant data has been planned to be shared with other researchers at this point since this is a feasibility study with only 40 participants

REFERENCES:
- [Derived] Ladha KS, Lee J, Mattina GF, Pazmino-Canizares J, Wijeysundera DN, Gholamali Nezhad F, Philip K, Tassone VK, Adamsahib F, Bhat V; SMILE Study Investigators. Sustained Mood Improvement with Laughing Gas Exposure (SMILE): Study protocol for a randomized placebo-controlled pilot trial of nitrous oxide for treatment-resistant depression. PLoS One. 2024 Jan 19;19(1):e0297330. doi: 10.1371/journal.pone.0297330. eCollection 2024. PMID 38241247